CLINICAL TRIAL: NCT04191447
Title: Multicenter, Randomized, Double-blind, Double-dummy, National, Phase III Clinical Trial to Evaluate the Efficacy and Safety of Flamboyant 200/12 Association in the Treatment of Adults With Severe Asthma .
Brief Title: Efficacy and Safety of Flamboyant 200/12 Association in the Treatment of Adults With Severe Asthma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EMS0319 - FLAMBOYANT200/12
Record Dates: First submitted 2019-12-05; First posted 2019-12-09 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind and double-dummy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FLAMBOYANT 200/12 (Experimental): The study is double-dummy. Thus, the participant must inhale 2 (two) capsules twice a day (12/12h), as follow:
  1 Flamboyant 200/12 capsule
  1 Budesonide/formoterol Placebo capsule.
  Interventions: Drug: Flamboyant 200/12; Other: Budesonide / Formoterol 400/12 Placebo
- Budesonide/formoterol 400/12 (Active Comparator): The study is double-dummy. Thus, the participant must inhale 2 (two) capsules twice a day (12/12h), as follow:
  1 Budesonide/formoterol 400/12 capsule
  1 Flamboyant 200/12 Placebo capsule.
  Interventions: Drug: Budesonide / Formoterol 400/12; Other: Flamboyant 200/12 Placebo

INTERVENTIONS:
Drug: Flamboyant 200/12 — Flamboyant 200/12 capsule
  Arms: FLAMBOYANT 200/12
Drug: Budesonide / Formoterol 400/12 — Budesonide / Formoterol 400/12 capsule
  Arms: Budesonide/formoterol 400/12
Other: Flamboyant 200/12 Placebo — Flamboyant 200/12 Placebo capsule
  Arms: Budesonide/formoterol 400/12
Other: Budesonide / Formoterol 400/12 Placebo — Budesonide / Formoterol 400/12 Placebo capsule
  Arms: FLAMBOYANT 200/12

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Flamboyant 200/12 association in adults with asthma.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the informed consent forms;
* Participants aged 18 years or more;
* Diagnosis of uncontrolled severe asthma;
* Participants with Forced expiratory volume in 1 second (FEV1) > 60% of predicted;

Exclusion Criteria:

* Any clinical and laboratory findings that, in the judgment of the investigator, may interfere with the safety of research participants;
* Known hypersensitivity to the formula components used during the clinical trial;
* History of alcohol and/or substance abuse within 12 months prior to Screening Visit.
* Current smoking or smoking history equivalent to "10 pack years"
* Participants with untreated oral candidiasis;
* Pulmonary disease history (e.g., chronic obstructive pulmonary disease [COPD], cystic fibrosis, bronchiectasis, tuberculosis);
* Participants with a history of acute asthma exacerbation, respiratory tract infection or hospitalization for asthma in the last 4 weeks;
* Known HIV-positive status or active hepatitis B or C virus test result
* Participants with current evidence or history of uncontrolled coronary artery disease, congestive heart failure, myocardial infarction or cardiac arrhythmia;
* Participants with a current medical history of cancer and/or cancer treatment in the last 5 years;
* Participants using medications that would have an effect on bronchospasm and / or lung function.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2022-07-22 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Forced expiratory volume in 1 second (FEV1), obtained through espirometry. | 12 weeks

SECONDARY OUTCOMES:
Incidence and severity of adverse events recorded during the study. | 14 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- IMC Tatuí, Tatuí, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162